CLINICAL TRIAL: NCT04876781
Title: Korean Post-marketing Surveillance for Xeljanz XR (Registered)
Brief Title: Korean Post-marketing Surveillance for Xeljanz XR
Acronym: XRPMS
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921369; NCT04876781 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-04-20; First posted 2021-05-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Active Moderate to Severe Rheumatoid Arthritis; Active Ankylosing Spondylitis; Active Psoriatic Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tofacitinib XR — Tofacitinib XR 11mg

SUMMARY:
Xeljanz XR extended-release tablets 11 mg (Tofacitinib citrate) is a drug subject to the risk management plan in accordance with Article 4-1-11 of the "Regulation on Safety of Medicinal Products, etc." in Korea. As part of additional pharmacovigilance activity, this Post-marketing Surveillance (PMS) was planned to evaluate safety and effectiveness of Xeljanz XR under routine clinical practice. At least 200 patients with Rheumatoid Arthritis, Psoriatic Arthritis, or Ankylosing Spondylitis who were treated with Xeljanz XR will be enrolled about four years.

DETAILED DESCRIPTION:
This is a open-label, non-comparative, non-interventional, prospective, and multi-center study to further evaluate the safety and effectiveness of Xeljianz XR in routine clinical practice in Korea.

Safety is the primary interest of this study, which will be assessed based on adverse events (AEs) that occur during the 6 months from the first dose of Xeljanz XR. The efficacy endpoints will be the modified Disease Activity Score using 28 joint counts (DAS28) change from baseline, European League Against Rheumatism (EULAR) response, and American College of Rheumatology 20% improvement criteria (ACR20) response after treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Xeljanz® XR is administered according to indications on the approved labeling

   * Treatment of moderate to severe active RA in adult patients (18 years of age or older) who have had an inadequate response or are intolerant to methotrexate
   * In combination with methotrexate, treatment of active psoriatic arthritis (PsA) in adult patients (18 years of age or older) who have had an inadequate response or who have been intolerant to a prior DMARD therapy.
   * Treatment of active ankylosing spondylitis (AS) in adult patients (18 years of age or older) who have responded inadequately to conventional therapy
   * In the following patients, Xeljanz® XR should be used only for patients who have had an inadequate response or are intolerant to the existing treatment.

   A. Patients aged 65 or older B. Cardiovascular high-risk patients C. Patients at risk for malignancy
2. Patients who have previously been given Xeljanz 5mg, who have changed Xeljanz® XR, are also eligible for registration in the study
3. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Patients with a history of hypersensitivity to any ingredients of this product.
2. Patients with serious infection (sepsis, etc.) or active infection including localized infection.
3. Patients with active tuberculosis.
4. Patients with severe hepatic function disorder.
5. Patients with an absolute neutrophil count (ANC) <1,000 cells/mm3. *
6. Patients with a lymphocyte count <500 cells/mm3. *
7. Patients with a hemoglobin level <9 g/dL. *
8. Pregnant or possibly pregnant women. * Do not initiate Xeljanz XR in the following cases: ANC; absolute neutrophil count <1,000 cells/mm3 ALC; absolute lymphocyte count <500 cells/mm3 Hemoglobin<9 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects administered with Xeljanz XR as a part of routine treatment who comply with the local labeling.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (AEs) | Maximum of 52 weeks from the time of initial administration of Xeljanz XR
  AE is any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to end of this PMS after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Xeljanz XR was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.

SECONDARY OUTCOMES:
Change from baseline in Disease Activity Score based on 28-joints Count (DAS28) | Baseline, 52 weeks after treatment or within 30 days after last dose of medicinal product
  DAS28, a modified version of the original Disease Activity Score (DAS), is a quantitative measure of disease activity used to monitor the treatment of RA.
Percentage of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28 | Baseline, 52 weeks after treatment or within 30 days after last dose of medicinal product
  The Disease Activity Score Based on 28-joints Count based (DAS28-based) EULAR response criteria is used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached.
Number of Participants With an American College of Rheumatology 20% (ACR20) Response | Baseline, 52 weeks after treatment or within 30 days after last dose of medicinal product
  ACR20 response: greater than or equal to (≥) 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Assessment of Ankylosing Spondylitis response (ASAS20) | Baseline, 52 weeks after treatment or within 30 days after last dose of medicinal product
  The ASAS Response Criteria (ASAS 20) is defined as an improvement of at least 20% and an absolute improvement of at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function (BASFI), and Inflammation (last 2 questions of BASDAI).
Changes from baseline in the number of tender joints and swollen joints | Baseline, 52 weeks after treatment or within 30 days after last dose of medicinal product
  The number of tender joints and swollen joints, which are the specific components of the ACR20 response, are measured. The improvement from baseline after treatment is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921369